CLINICAL TRIAL: NCT06602193
Title: A Phase 2a, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Pharmacodynamic Effects of BIIB122 in Participants With LRRK2-Associated Parkinson's Disease (LRRK2-PD)
Brief Title: Safety and Pharmacodynamic Effects of BIIB122 in Participants With LRRK2-Associated Parkinson's Disease (LRRK2-PD)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Denali Therapeutics Inc. (Industry)
Collaborators: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DNLI-C-0009
Record Dates: First submitted 2024-09-16; First posted 2024-09-19 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-07

CONDITIONS: Parkinson Disease
Keywords: LRRK2; Movement Disorders
MeSH Terms: conditions — Parkinson Disease; Movement Disorders | interventions — DNL151

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BIIB122 225 mg (Experimental): Oral 225 mg dose, once daily (QD)
  Interventions: Drug: BIIB122 225 mg
- BIIB122 Matching Placebo (Placebo Comparator): Oral BIIB122 matching placebo, once daily (QD)
  Interventions: Other: BIIB122-Matching Placebo

INTERVENTIONS:
Drug: BIIB122 225 mg — Administered as specified in the treatment arm
  Other Names: DNL151
  Arms: BIIB122 225 mg
Other: BIIB122-Matching Placebo — Administered as specified in the treatment arm
  Arms: BIIB122 Matching Placebo

SUMMARY:
This Phase 2a, multicenter, randomized, 12-week double-blind, placebo-controlled, parallel-group study, followed by an OLE, is designed to evaluate the safety, tolerability, and pharmacodynamic effects of BIIB122 in participants with LRRK2-PD. LRRK2-PD is defined as Parkinson's Disease (PD) in individuals who are heterozygous or homozygous carriers of a pathogenic LRRK2 variant that increases LRRK2 kinase activity.

ELIGIBILITY:
Inclusion Criteria:

* For heterozygous pathogenic LRRK2 mutation carriers: ≥ 30 to ≤ 80 years
* For homozygous pathogenic LRRK2 mutation carriers: ≥ 30 years
* Have screening genetic test results verifying the presence of a pathogenic LRRK2 variant.
* Have a clinical diagnosis of PD meeting the Movement Disorder Society Clinical Diagnostic Criteria.

Exclusion Criteria:

* Have a history of any clinically significant neurological disorder other than PD, including, but not limited to, stroke and dementia, in the opinion of the investigator, within 5 years of the screening visit.
* Have clinical evidence of atypical parkinsonism (eg, multiple-system atrophy or progressive supranuclear palsy) or evidence of drug-induced parkinsonism.
* Have previously participated or are currently participating in the BIIB122 LUMA study (Study 283PD201).
* Have previously participated or are currently participating in a gene therapy study for PD.
* Have a history of brain surgical intervention for PD (eg, deep-brain stimulation, pallidotomy).
* Have any physical condition that may confound the motor assessment (MDS-UPDRS) over time (eg, severe arthritis, severe dyskinesias, traumatic injuries with permanent physical disability).
* Abnormal vitals including Blood Pressure, Heart Rate, or Body Temperature
* Have abnormal PFT results at screening

Note: Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) with BIIB122 compared with placebo over the 12-week double-blind period | 12 weeks

SECONDARY OUTCOMES:
Change from baseline in whole-blood pS935 LRRK2 with BIIB122 compared with placebo at Week 12 | 12 weeks
Change from baseline in urine BMP with BIIB122 compared with placebo at Week 12 | 12 weeks

OTHER OUTCOMES:
Incidence of TEAEs and SAEs during the OLE period | 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Danna Jennings, MD, Study Director — Denali Therapeutics
Locations (16):
- United States (7):
  - Cedars-Sinai Department of Neurology, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - Parkinson's Disease and Movement Disorders Center, Boca Raton, Florida
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Ichan School of Medicine at Mount Sinai/Beth Israel Downtown-Movement Disorder Center, New York, New York
  - Evergreen Health Laboratory, Kirkland, Washington
  - Inland Northwest Research, Spokane, Washington
- Germany (3):
  - Technische Universität Dresden, Dresden
  - University of Lübeck, Lübeck
  - University Hospital Tübingen, Tübingen
- Spain (6):
  - Hospital Universitari General de Catalunya, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Donostia, Donostia / San Sebastian
  - Universitary Hospital La Princesa, Madrid
  - IDIVAL/University Hospital Marques de Valdecilla, Santander
  - Hospital Universitario Virgen del Rocio, Seville

IPD SHARING:
Plan to Share IPD: No